CLINICAL TRIAL: NCT04081480
Title: Pharmacokinetics of a New Paediatric Formulation of Valacyclovir Used for Prophylaxis and Treatment of Varicella Zoster Virus (VZV) and Herpes Simplex Virus (HSV) Infections in Children, Phase II (VALID II)
Brief Title: Pharmacokinetics of Valacyclovir Oral Solution in Children
Acronym: VALID2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed positive results, it was difficult to include patients and also the fact that the grant for this project has ended, we have decided to complete the study before we had included the total number of 16 patients.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VALID2
Record Dates: First submitted 2019-07-16; First posted 2019-09-09 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Herpes Simplex Virus Infection; Varicella Zoster Virus Infection
MeSH Terms: conditions — Herpes Simplex; Varicella Zoster Virus Infection | interventions — Valacyclovir

STUDY DESIGN:
Intervention Model Description: Intervention is pharmacokinetic (PK) curve collection in children, two age groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Valacyclovir oral solution (Other): Valacyclovir oral solution as administered in standard of care. Dosage: 10 mg/kg BID for children weighing less than 40 kg and 500 mg BID for children weighing 40 kg or more.
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir — PK curve collection to determine acyclovir exposure after administration of valacyclovir oral solution

SUMMARY:
Valacyclovir has replaced acyclovir in many clinical scenarios. Pharmacokinetic data support the use of oral valacyclovir in children, but practical problems exist in children having to take adult-dose tablets. A formulation with acceptable palatability, good pharmaceutical quality and possibility of flexible dosing is developed. Pharmacokinetic data of this formulation is missing.

The present study investigates the pharmacokinetics of valacyclovir oral solution in children by determine the area under the curve (AUC0-12), time above critical concentration (Ccrit), Cmax and Tmax of acyclovir.

Secondary, the safety profile of a single dose of valacyclovir oral solution will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in the age of 2-12 years.
* Subject has an indication for (val)acyclovir prophylaxis and are planned to receive valacyclovir oral solution.
* Subject is managed with a central venous catheter (CVC/Port-a-Cath).
* Subject's parents have signed the Informed Consent Form prior to screening evaluations.
* Subject is willing to participate after study procedures are explained in comprehensible language for the child.

Exclusion Criteria:

* Severe anemia (<6.0 mmol/L).
* Full dose has not been taken.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve | 12 hours
  Acyclovir area under the curve (12h)
Cmax | 12 hours
  Maximum concentration of aciclovir
Tmax | 12 hours
  Time to reach maximum concentration of aciclovir

SECONDARY OUTCOMES:
Number of adverse events | 1 day
  Number of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Prinses Maxima Centrum voor kinderoncologie, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No